CLINICAL TRIAL: NCT06784648
Title: An Open-Label, Multicentre Phase 1B/2A Clinical Trial of BI-1607, an Fc-Engineered Monoclonal Antibody to FcγRIIB (CD32B) in Combination With Ipilimumab and Pembrolizumab in Participants With Unresectable or Metastatic Melanoma
Brief Title: Different Doses of BI-1607 in Combination With Pembrolizumab and Ipilimumab, in Participants With Unresectable or Metastatic Melanoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioInvent International AB (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-BI-1607-02; 2024-512670-10 (EudraCT Number); KEYNOTE-G05 (Other: Merck Sharp & Dohme LLC); MK-3475-G05 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2024-12-16; First posted 2025-01-20 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Melanoma Metastatic; Melanoma of Skin; Melanoma BRAF V600E/K Mutated; Melanoma Recurrent; Melanoma Stage III or IV; Melanoma; Melanoma Negative for bRAF; Melanoma Negative for nRAS; Melanomas; Uveal Melanoma, Metastatic
Keywords: anti-CTLA-4; anti-PD-1; resistant anti-PD-1; progressed on treatment with an anti-PD-1/L1; metastatic
MeSH Terms: conditions — Melanoma; Uveal Melanoma; Neoplasm Metastasis | interventions — pembrolizumab; Ipilimumab; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination of BI-1607, Ipilimumab and pembrolizumab (Experimental): In each cohort in phase Ib BI-1607 will be given with ipilimumab in 3-week cycles for 4 cycles in combination with pembrolizumab (KEYTRUDA) from cycle 3 for up to 2 years from start of treatment.
  In the phase 2 pembrolizumab (KEYTRUDA) will be given in combination with BI-1607 and ipilimumab in 3-week cycles for 4 cycles then a pembrolizumab (KEYTRUDA) monotherapy will be provided from cycle 5 for up to 2 years from start of treatment.
  Interventions: Biological: pembrolizumab (KEYTRUDA®); Biological: BI-1607; Biological: Ipilimumab (YervoyTM, 50 mg/10 mL solution)

INTERVENTIONS:
Biological: pembrolizumab (KEYTRUDA®) — fixed dose 200mg
Biological: BI-1607 — Each cohorts will receive either 350mg or 700mg per cycle for 4 cycles
Biological: Ipilimumab (YervoyTM, 50 mg/10 mL solution) — Each cohort will receive either 1mg/kg or 3mg/kg for 4 cycles

SUMMARY:
Why the research is needed: Researchers are looking for a better way to treat melanoma that has spread or cannot be removed surgically. Melanoma is a type of skin cancer that starts in melanocytes, the cells that make the pigment that gives skin its color. In people with cancer, the body cannot control the growth of cells, which can come together to form tumors. This trial's new treatment is called BI-1607. BI-1607 is designed to work by improving the effectiveness of other targeted therapies already used for melanoma treatment; ipilimumab and pembrolizumab. BI-1607 will improve the ability of these two treatments to help the body's defense system to destroy cancer cells.

DETAILED DESCRIPTION:
Trial Participants: This trial will include an estimated number of 35 participants with melanoma cancer who have not been helped by standard treatments.

The main purposes of this trial are :

1. To learn about the safety and tolerability of BI1607 when received in combination with ipilimumab and pembrolizumab,
2. To determine the best dose (quantity) of both BI-1607 and ipilimumab when combined with pembrolizumab, and
3. To see if this triple combination therapy of BI-1607/ipilimumab/ pembrolizumab is more effective.

To investigate this, the researchers will study:

* what medical problems can happen during the trial, whether there are changes in the participants' health, how many participants reduce their dose of treatment or stop treatment for a period during the trial, and how many participants have medical problems that cause them to stop their trial treatment early.
* how many participants have dose-limiting toxicities (also called "DLTs", which are medical problems severe enough to stop the trial doctors from increasing a treatment dose in the next group of participants).

  2. The researchers will also study the following additional questions in this trial:
* how BI-1607 acts in the body when received with ipilimumab/pembrolizumab.
* whether the triple combination at varying doses of BI-1607 and ipilimumab acts in the participants' bodies as expected and has a desired effect on certain proteins in the participants' immune systems.
* the number of participants who produce "antibodies" against BI-1607 and tolerability. Antibodies are proteins which are part of the immune system that help fight an infection. However, the body can produce antibodies against a treatment, which can stop the treatment from working properly.
* how many participants' tumors shrink after receiving BI-1607 in combination with ipilimumab/pembrolizumab, and how long do their tumors shrink before their melanoma get worse or they pass away.

What is planned to happen during this trial: The participants are planned to be in this trial for a maximum of 25.5 months. This trial started end of 2024 and is planned to end in 2028.

This trial will have 2 parts, called Phase 1 and Phase 2.

In Phase 1, at least 15 participants will receive BI-1607 and ipilimumab once every three weeks over four treatment time points, i.e., 12 weeks. Pembrolizumab will be added to the combination treatment at the third and fourth treatment. If the participant continues in the trial thereafter, pembrolizumab will be administered alone every third week from the fifth week onwards, up to a total of 35 treatments or approximately 2 years. This phase 1 will likely contain 4 groups of participants receiving different dose levels of treatments. After the participants in the first dose group have received their first treatments, the Sponsor, in collaboration with researchers, decides if this dose is safe, and the dose will be increased in the next group of participants.

In Phase 2, approximately 20 participants will receive BI-1607 at the selected dose that the Sponsor and researchers decide is safe during Phase 1. BI-1607 will be administered once every three weeks in combination with both ipilimumab and pembrolizumab over four treatment time points, i.e., 12 weeks. Thereafter, pembrolizumab will be administered alone every third week, up to a total of 35 treatments or approximately 2 years.

In both phases, the treatments will be administered via an "IV infusion" in which an IV line is inserted into a vein usually in the arm. The treatments will be dosed in milligrams, also called "mg". The lowest dose of BI-1607 will be 350 mg, and the highest possible dose will be 700 mg. Ipilimumab will be given to participants at a dose of 1 mg/kg body weight or 3 mg/kg. The dose of pembrolizumab will be 200 mg.

Throughout the trial, the researchers will check the participants' health and any medical problems, ask about any medications they are receiving, take blood, tumor, and urine samples, and scan their tumors. The researchers will do these tests to learn how safe BI-1607 is in combination with ipilimumab/pembrolizumab, how the drug acts in the body, and how the treatment affects the participants' tumors.

Benefits of this trial: There is no guarantee that the participants will receive any benefit from participating in this trial. However, their participation may help other people who have melanoma receive better care in the future.

Risks of this trial: Participant safety is the most important factor in clinical trials. However, it cannot be guaranteed that the participants will not have medical problems during this trial. The clinical researcher will determine if the participant should no longer take part in the study if the results show the treatment doses are not safe. The Sponsor, Ethics Committee, or Regulatory Authority may also decide to stop the study at any time for any reason.

ELIGIBILITY:
Inclusion Criteria:

1. Is willing and able to provide written informed consent for the trial.
2. Is ≥ 18 years of age on the day of signing informed consent.
3. Has histologically confirmed advanced melanoma (unresectable or metastatic melanoma) with established disease progression.
4. Participants must have progressed on treatment with an anti-PD-1/L1 mAb. Subjects with uveal melanoma are not required to have received any prior anti-PD-1/L1 treatment. PD-1 treatment progression is defined by meeting all of the following criteria:

   1. Has received at least 2 doses of an approved anti-PD-1/L1 mAb.
   2. Has demonstrated disease progression after anti PD-1/L1 as defined by RECIST v1.1.

      The initial evidence of disease progression is to be confirmed by a second assessment no less than four weeks from the date of the first documented disease progression, in the absence of rapid clinical progression.
   3. Progressive disease has been documented within 12 weeks from the last dose of anti-PD-1/L1 mAb.
5. Participants may have received previous treatment with BRAF inhibitors alone or in combination with mitogen extracellular kinase (MEK) inhibitors.
6. Has at least 1 measurable disease lesion as defined by RECIST v1.1 criteria.
7. Must be willing to provide tumour biopsies as specified in the schedule of assessments (SoA) unless otherwise discussed and agreed with the Sponsor in case a biopsy cannot be taken for a medical/safety reason.
8. Has a life expectancy of ≥ 12 weeks.
9. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
10. Has adequate organ function as confirmed by laboratory values
11. Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to enrolment.
12. Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at Screening.

Exclusion Criteria:

1. Has previously been treated with an anti-CTLA-4 mAb or anti-LAG3 mAb (anti-Lymphocyte Activation Gene 3).
2. Has received any prior immunotherapy and was discontinued from that treatment due to a Grade 3 or higher irAE (except endocrine disorders that can be treated with replacement therapy) or was discontinued from that treatment due to Grade 2 myocarditis or recurrent Grade 2 pneumonitis.
3. Has received the following:

   1. Chemotherapy or small molecule products within 4 weeks of first dose of BI-1607.
   2. Radiotherapy within 2 weeks of first dose of BI-1607, or has radiation-related toxicities, requiring corticosteroids. Participants who have previously had radiation pneumonitis are not allowed.
   3. Immunotherapy or biological anti-cancer therapy or an investigational agent or an investigational device within 4 weeks prior to the first dose of BI-1607.
4. Has not recovered from all AEs due to previous therapies to ≤ Grade 1 or baseline.
5. Has had major surgery from which the participant has not yet recovered or is scheduled to have major surgery < 28 days prior to the first dose of trial intervention.
6. Has received a live or live-attenuated vaccine within 30 days prior to the first dose of trial intervention.
7. Is participating or planning to participate in another interventional clinical trial or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to first dose of trial intervention.
8. Has history of allogeneic tissue/solid organ transplant.
9. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of trial intervention .
10. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
11. Has known active CNS metastases and/or carcinomatous meningitis.
12. Has severe hypersensitivity to (≥ Grade 3) to pembrolizumab and/or any of its excipients. Has known or suspected hypersensitivity to BI-1607, ipilimumab or any of their excipients. Previous isolated infusion related reactions (IRRs) are not to be considered a reason for exclusion unless Grade 4 in severity.
13. Has an active autoimmune disease that has required systemic treatment in past 2 years.
14. Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
15. Is at high medical risk because of non-malignant systemic disease including severe active infections on treatment with antibiotics, antifungals, or antivirals.
16. Has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority.
17. Has cardiac or renal amyloid light-chain amyloidosis.
18. Is a female participant and has the possibility to become pregnant (or already pregnant or lactating/breastfeeding). However, those female participants who have a negative serum or urine pregnancy test before enrolment and agree to use a highly effective method of birth control for 4 weeks before entering the trial, during the trial, and for 12 months after last dose of BI-1607 OR 4 months after the last dose of pembrolizumab, whichever is later are considered eligible.
19. Is a male participant with partner(s) of childbearing potential (unless he agrees to use a barrier method of contraception with the female partner(s) who are using one highly effective method of contraception during the trial and for 12 months after completing treatment).
20. Has uncontrolled or significant cardiovascular disease
21. Has a history or there is current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or in the opinion of the treating Investigator is not in the best interest of the participant to participate.
22. Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | end of Cycle 4 (each cycle is 21 days)
  The frequency and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) will be assessed.
Safety and tolerability | end of Cycle 4 (each cycle is 21 days)
  The frequency of dose interruptions, dose modifications and trial intervention discontinuations will be evaluated.
Safety and tolerability | end of Cycle 4 (each cycle is 21 days)
  Changes of body temperature following the infusions will be assessed.
Safety and tolerability | end of Cycle 4 (each cycle is 21 days)
  ECG will be performed and the QTc will be used to assess the cardiac safety.
Safety and tolerability | end of Cycle 4 (each cycle is 21 days)
  Changes in concentrations of hematology laboratory parameters (platlet count, red blood cells count, white blood cells count) will be assessed.
Safety and tolerability | end of Cycle 4 (each cycle is 21 days)
  Changes in blood pressure following the infusions will be assessed.
Safety and tolerability | end of Cycle 4 (each cycle is 21 days)
  Changes in respiration rate following the infusions will be assessed.
Safety and tolerability | end of Cycle 4 (each cycle is 21 days)
  Changes in pulse rate following the infusions will be assessed.
Recommended doses for the expansion cohort | End of Cycle 3 (each cycle is 21 days)
  During phase 1b, to determine the recommended doses for expansion of BI-1607 and ipilimumab in combination with pembrolizumab.
Efficacy | Through study completion, a maximum of 2 years
  Phase 2a: The best tumour response rate (according to Response Evaluation Criteria in Solid Tumour (RECIST) v.1.1 and immune RECIST (iRECIST)) will be used to assess the efficacy.
Efficacy | Through study completion, a maximum of 2 years
  Phase 2a: The objective response rate (according to Response Evaluation Criteria in Solid Tumour (RECIST) v.1.1 and immune RECIST (iRECIST)) will be used to assess the efficacy.
Efficacy | Through study completion, a maximum of 2 years
  Phase 2a: The progression-free survival (PFS) measured in months will be used to assess the efficacy.
Efficacy | Through study completion, a maximum of 2 years
  Phase 2a: The time to response measured in months will be used to assess the efficacy.
Efficacy | Through study completion, a maximum of 2 years
  Phase 2a: The duration of response (DoR) measured in months will be used to assess the efficacy.
Efficacy | Through study completion, a maximum of 2 years
  Phase 2a: The overall survival (OS) measured in months will be used to assess the efficacy.
Safety and tolerability | end of Cycle 4 (each cycle is 21 days)
  Changes in concentrations of clinical chemistry concentrations in blood (haemoglobin, creatinin, albumin, blood urea nitrogen, potassium, sodium, calcium, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, bilirubin, total proteins and phosphate) will be assessed.

SECONDARY OUTCOMES:
Pharmacokinetics profile of BI-1607 | end of Cycle 4 (each cycle is 21 days)
  The PK parameters assessed will include area under the concentration time curve (AUC).
Pharmacokinetics profile of BI-1607 | end of Cycle 4 (each cycle is 21 days)
  The PK parameters assessed will include the maximum concentration (Cmax).
Pharmacokinetics profile of BI-1607 | end of Cycle 4 (each cycle is 21 days)
  The PK parameters assessed will include the area under the plasma concentration versus time curve (AUC).
Pharmacokinetics profile of BI-1607 | end of Cycle 4 (each cycle is 21 days)
  The PK parameters assessed will include the terminal half-life (t1/2).
Immunogenicity of BI-1607 when administered in combination with ipilimumab and pembrolizumab | end of Cycle 4 (each cycle is 21 days)
  To assess the incidence and titre of antidrug antibodies to BI-1607 in blood serum

OTHER OUTCOMES:
Expression levels of Fc receptors, and other immunological and melanoma disease markers | end of Cycle 4 (each cycle is 21 days)
  To investigate the mRNA expression levels of Fc receptors, including FcγRIIB (protein and/or nucleic acids) and other immunological and melanoma disease markers (e.g., PD-1, LDH), and to study a potential correlation of levels of expression with clinical responses.
Genetic background of participants with respect to FcgR | First day of treatment
  To investigate the genetic variants of participants with respect to FcgR isoforms and explore a potential correlation of the genetic background with clinical responses.

CONTACTS AND LOCATIONS:
Locations (9):
- Germany (4):
  - Charité - Universitatsmedizin Berlin, Berlin
  - University Hospital Essen, Essen
  - University Hospital Heidelberg, Heidelberg
  - University Medical Center Mannheim, Ruprecht-Karl University of Heidelberg and Clinical Cooperation Unit Dermato-Oncology(G300) German Cancer Research Center(DKFZ), Mannheim
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - University Hospital 12 de Octubre, Madrid
- United Kingdom (3):
  - Sarah Cannon Research Institute UK, London, Greater London
  - Velindre Cancer Centre, Cardiff, Wales
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
All information concerning the product as well as any matter concerning the operation of the Sponsor, such as clinical indications for the drug, its formula, methods of manufacture and other scientific data relating to it, that have been provided by the Sponsor and are unpublished, are confidential and must remain the sole property of the Sponsor. The Investigator will agree to use the information only for the purposes of carrying out this study and for no other purpose unless prior written permission from the Sponsor is obtained.
Supporting Information: Study Protocol, CSR
Time Frame: 1 year after the last patient last visit.
Access Criteria: Abbreviated CSR published online